CLINICAL TRIAL: NCT03716804
Title: Introduction of Nitrofurantoin in Place of Ciprofloxacin in Patients of Uncomplicated Urinary Tract Infection: a Controlled Clinical Trial to Establish the Relationship Between Revival and Associated Shift in Sensitivity Pattern of the Causative Microbes
Brief Title: Establish the Relationship Between Shift in Prescribing Pattern and Associated Shift in Sensitivity Pattern of Causative Microbes in UTI Patients in a Closed Community
Acronym: UTI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Dr. Sabiha Mahboob, Resident, Phase B, Pharmacology, BSMMU, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: BSMMU/2018/4643
Record Dates: First submitted 2018-10-17; First posted 2018-10-23 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Uncomplicated Urinary Tract Infection; Antibiotic Resistant Infection

STUDY DESIGN:
Intervention Model Description: Parallel assignment Intervention group: Educational intervention to prescribers and Medicine-Tab Nitrofurantoin (100 mg, 2 times daily for 7 days) to the patients.
  Control group: No educational intervention to the prescribers and Medicine- of personal choice of physician(Tablet Ciprofloxacin, 500 mg/Tablet Cef 3, 200 mg/Tab Cefuroxime, 250 mg) to the patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Intervention:
  To the prescribers- Educational intervention about guideline and present sensitivity trend.
  To the Patients- Tablet Nitrofurantoin(100 mg), two times daily at 12 hours interval for 7 days.
  Interventions: Drug: Tablet Nitrofurantoin
- Control Group (Active Comparator): Intervention:
  To the Patients- Tablet Ciprofloxacin, 500 mg or,Tablet Cefixime 200 mg or,Tablet Cefuroxime 250 mg (According to physician's personal choice).
  Interventions: Drug: Tablet Ciprofloxacin/ Tablet Cefixime/ Tablet Cefuroxime

INTERVENTIONS:
Drug: Tablet Nitrofurantoin — Tablet Nitrofurantoin (100 mg), two times daily in 12 hours interval for 7 days
  Arms: Intervention group
Drug: Tablet Ciprofloxacin/ Tablet Cefixime/ Tablet Cefuroxime — Tablet Ciprofloxacin (500 mg), two times daily in 12 hours interval for 7 days or, Tablet Cefixime (200 mg), two times daily in 12 hours interval for 7 days or, Tablet Cefuroxime (250 mg), two times daily in 12 hours interval for 7 days
  Arms: Control Group

SUMMARY:
To establish a relationship between changed prescribing pattern and associated shift in sensitivity trend of causative microbes in patients of uncomplicated urinary tract infection in a closed community

DETAILED DESCRIPTION:
Antibiotic resistance has become a startling issue in last two decades. Many strategies are being followed to combat antibiotic resistance; revival of older, effective antibiotics is one of those approaches. Urinary tract infection is one of the most common indication for which antibiotics are prescribed. Despite having published guidelines in urinary tract infection, studies show that there is wide variability in prescription. The proposed study is designed to reinforce the guideline among a group of prescribers and evaluate the associated shift in sensitivity pattern of common urinary pathogens. This study will be a double center, controlled clinical trial. In this study, the prescribers in intervention arm will be given educational intervention and in control arm no intervention will be given. When a patient is diagnosed as a case of uncomplicated urinary tract infection clinically in intervention arm, after fulfilling the study criteria the patient will be enrolled in the study. Prescription data will be collected on daily basis and sensitivity data will be collected monthly. Clinical outcome of the patients enrolled in the study will be measured over telephone, after completion of their treatment. Sensitivity pattern will be analysed monthly after collection of sensitivity data from the laboratory affiliated with the hospital. All these data will be compiled and analysed at the end of the study. In control arm, prescription data will be collected fortnightly and sensitivity data will be collected monthly. All these data will be compiled and analysed at the end of the study. After approval from the institutional review board (IRB), enrolled patient will be informed about the intervention and the study.Informed written consent will be taken from all the patients, who will take part in the study willingly. Patient's anonymity will be maintained and will be used for study purpose only.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed uncomplicated urinary tract infection
* Patient agreed to participate in the study signing an informed written consent

Exclusion Criteria:

* Known hypersensitivity to Nitrofurantoin
* Known Case of Diabetes mellitus, Hypertension, glucose-6-phosphate dehydrogenase deficiency
* Suspected complicated or recurrent UTI
* Elderly Patients of 65 years or more
* Neonates ang pregnant women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2018-06-06 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Shift in sensitivity pattern of microorganisms in urinary pathogens | Upto 6 months
  After shift of prescription from Ciprofloxacin to Nitrofurantoin in patients of UTI, the associated shift in sensitivity pattern of causative microbes will be ruled out by analysing the urine culture-sensitivity data from affiliated pathology lab

SECONDARY OUTCOMES:
Non-inferiority of the drug | 7 days after start of the antibiotic therapy
  Clinical outcome of the patients will be measured over Phone interview after completion of antibiotic treatment.
  Indicator:Total patients cured after the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Md. Sayedur Rahman, MBBS,Mphil,FCPS, Study Chair — Head of the Department, Department of Pharmacology, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Locations (1):
- Combined Military Hosptal, Dhaka, Dhaka, Bangladesh